CLINICAL TRIAL: NCT06626711
Title: Effect of Propofol and Sevoflurane Anesthesia on HSP70 Expression in Tumor Cells A Prospective, Single-center, Pilot, Randomized Study
Brief Title: Effect of Propofol and Sevoflurane Anesthesia on HSP70 Expression in Tumor Cells
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Collaborators: Institute of Cytology of the Russian Academy of Sciences (Unknown); The Russian Science Foundation (Unknown)
Responsible Party: Principal Investigator, Efremov Sergey, Deputy director for science, Saint-Petersburg state university hospital, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-25-00078
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia; Cancer Recurrence; Cancer
Keywords: Cancer; Anesthesia; Sevoflurane; Propofol
MeSH Terms: conditions — Neoplasms | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol-based total venous anesthesia group (Experimental): These patients will receive total venous anethesia where propofol is used as a hypnotic drug.
  Interventions: Drug: Propofol
- Sevoflurane-based inhalational anesthesia group (Experimental): These patients will receive inhalational anethesia where sevoflurane is used as a hypnotic drug.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Propofol as a part of total venous anesthesia
  Arms: Propofol-based total venous anesthesia group
Drug: Sevoflurane — Sevoflurane as a part of intravenous anesthesia
  Arms: Sevoflurane-based inhalational anesthesia group

SUMMARY:
The goal of this clinical trial is to learn if sevoflurane-based inhalational anesthesia (s-IA) and propofol-based total intravenous anesthesia (p-TVA) have different effects on HSP70 expression in different types of tumour cells. The main questions it aims to answer are:

* if p-TVA/s-IA increase or suppress HSP70 expression in tumor cells in comparison with a pre-anesthesia level;
* does this change in HSP70 expression cause any difference in vital characteristics of tumor cells, such as proliferation, apoptosis, colony formation and migration.

Researchers will compare p-TVA with s-IA by ability of these types of anesthesia to change the HSP70 expression level and modulate HSP70-mediated effects in tumor cells.

Participants will:

* be randomly allocated to p-TVA or s-IA groups;
* donate 12 ml of blood before anesthesia induction and 12 ml after 2 hours of anesthesia.

The blood serum will be used to prepare cell medium. After exposure to this medium, cells from different tumor types will be investigated using cytological and molecular biological methods.

DETAILED DESCRIPTION:
This study will be conducted in adult cancer patients who undergo planned radical or palliative tumor resection and signed informed consent. Patients with diabetes mellitus, HIV, hepatitis B and C, as well as patients who undergo emergency surgery will not be included to the study. Patients will be randomly allocated to propofol-based TVA (p-TVA) and sevoflurane-based IA (s-IA) groups. After the collection of blood before the anesthesia induction and in 2 hours of anesthesia, probes will be centrifuged to prepare serum. Cell medium will contain 50% of blood serum. Different tumor cell lines (human lung adenocarcinoma A549, large cell lung carcinoma NCI-H460, human colorectal adenocarcinoma DLD1) will be exposed to the cell medium for 4 hours what corresponds to an approximate duration of anesthesia for oncology surgery. HSP70 expression level will be determined using SDS-PAGE (polyacrilamide gel electrophoresis) and Western-blot analysis (intracellular HSP70 content), ELISA of cell medium (extracellular HSP70 expression) and confocal microscopy.

The A549 cell line with stable knockdown of HSP70 developed by shRNA will be used to distinguish HSP70-based effects of cell medium from p-TVA and s-IA groups on vital characteristics of tumor cells, including proliferation (MTT assay), apoptosis (LDH cytotoxicity assay), colony formation and migration (the Wound healing assay).

Researchers will compare HSP70 expression levels and vital characteristics of tumor cells exposed to patient serum before and after each type of anesthesia, as well as p-TVA group with s-IA group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed malignant neoplasm
* Planned surgery for radical or palliative tumor resection
* Age over 18 years
* Signed informed consent

Exclusion Criteria:

* Diabetes mellitus type 2
* HIV, hepatitis B or C
* Emergency surgery
* Known or suspected allergy to studied drugs
* Other conditions when one of the types of anesthesia is more preferable (hemodynamic disorders, bronchial asthma etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
HSP70 expression in tumor cells in vitro | 24 hours after exposition with patients serum.
  Increased intracellular and extracellular HSP70 content in different types of tumor cells measured by SDS-PAGE/Western blotting and ELISA, respectively.

SECONDARY OUTCOMES:
LDG cytotoxicity | 24 hours after exposition with patients serum.
  Reduction of apoptosis mediated by HSP70 pathway in different types of tumor cells measured by LDG cytotoxicity assay using HSP70-knockdown cell line.
MTT test | 24 hours after exposition with patients serum.
  Increase in proliferation mediated by HSP70 pathway in different types of tumor cells measured by MTT assay using HSP70-knockdown cell line.
Wound healing test | 72 hours after exposition with patients serum.
  Increase in cell migration mediated by HSP70 pathway in different types of tumor cells measured by the Wound healing assay.
Cell colonies formation | 7 days after exposition with patients serum.
  Increase in ability to form colonies mediated by HSP70 pathway in different types of tumor cells evaluated by direct microscopy using HSP70-knockdown cell line.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01/10/2024 - 01/04/2025
Access Criteria: By reasonable request.